CLINICAL TRIAL: NCT04884022
Title: Effectiveness of Two Skeletally Anchored Force Mechanics for Correction of Skeletal Class II Malocclusion in Growing Patients (A Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Two Skeletally Anchored Force Mechanics for Skeletal Class II Correction in Growing Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yasmine Mohamed Sayed Mahmoud, clinical researcher, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anchored force mechanices
Record Dates: First submitted 2021-04-24; First posted 2021-05-12 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Miniplates in mandibular symphysis & infrazygomatic (Experimental)
  Interventions: Procedure: Miniplates in mandibular symphysis & infrazygomatic
- Miniplates in external oblique ridge & anterior maxillary region (Active Comparator)
  Interventions: Procedure: Miniplates in external oblique ridge & anterior maxillary region
- Growing skeletal Class II subjects (No Intervention)

INTERVENTIONS:
Procedure: Miniplates in mandibular symphysis & infrazygomatic — Fixed functional appliance (pushing orthopedic force) in conjunction with direct skeletal anchorage
  Arms: Miniplates in mandibular symphysis & infrazygomatic
Procedure: Miniplates in external oblique ridge & anterior maxillary region — Coil spring (pulling orthopedic force) in conjunction with direct skeletal anchorage
  Arms: Miniplates in external oblique ridge & anterior maxillary region

SUMMARY:
Patients with skeletal Class II malocclusion due to mandibular retrognathism will be recruited and randomly allocated to three equal groups. first group will be treated by pushing orthopedic force mechanics, second group will be treated by pulling orthopedic force mechanics, and third group will be observed for 9 months to detect the natural growth changes. Skeletal changes will be evaluated and the treatment changes will be compared with the natural growth changes. The study hypothesis is that use of direct bimaxillary miniplate anchorage in conjunction with fixed functional appliance (pushing orthopedic force) or closed coil spring (pulling orthopedic force) will induce statistically significant skeletal mandibular growth in comparison to natural mandibular growth changes.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be conducted to address the aim of the study. Thirty-nine growing patients with skeletal Class II malocclusion due to mandibular retrognathism will be recruited. The sample will be randomly allocated to three equal groups, each including thirteen subjects. Group A will be treated by pushing orthopedic force mechanics using fixed functional appliance (Sabbagh Advanced Repositioning Appliance) anchored to four miniplates (two miniplates inserted in the mandibular symphysis and two infrazygomatic miniplates), and Group B, will be treated by pulling orthopedic force mechanics using Class II springs (CS Class II correction device) anchored to four miniplates (two inserted in the mandibular posterior buccal segment and two inserted in the maxillary anterior segment). In both groups, the appliances will be removed after reaching an edge-to-edge incisor relationship or after 9 months, whichever happens first. A similar third group (Group C) will be observed for 9 months to detect the natural growth changes. Skeletal changes will be evaluated using pretreatment and posttreatment cone beam computed tomography scans (CBCT). The treatment changes will be compared with the natural growth changes observed in group C. Other variables will be also examined including, the dentoalveolar effects, the soft tissue profile, and the patient's acceptance to this treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age ranges from 11 years to 13 years.
* Skeletal Class II malocclusion with a deficient mandible (SNB ≤ 76°).
* Horizontal growth pattern (MP/SN ≤ 39°).
* Angle Class II division 1 malocclusion with at least 5 mm overjet.
* Mandibular arch crowding less than 5 mm.
* The patients have to be in the prepubertal growth stage (cervical maturational stage 3 or 4) when applying orthopedic force.
* Patients with good oral hygiene, and a healthy periodontal condition.

Exclusion Criteria:

* Patients who underwent previous orthodontic treatment.
* Patients with previous craniofacial surgeries, chronic diseases, syndromes, or growth problems that may affect bone.
* Any signs or symptoms of para-functional habits or previous history of temporomandibular disorders.
* Extracted or missing upper permanent teeth (except for third molars).

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
change in the effective mandibular length (Co-Gn) | at baseline and after treatment completion about 9 months
  Correction of the skeletal Class II relation. This outcome will be detected by measuring the mean change in the effective mandibular length (Co-Gn) and position on CBCT images from baseline data (T1) and after appliance removal (T2) and will be compared with the growth changes observed in the control group

SECONDARY OUTCOMES:
change in maxillary length (Co-A) | at baseline and after treatment completion about 9 months
  The effective maxillary length (Co-A) and position changes will be measured after and chin will be measured.
Changes in the soft tissue angle of convexity | at baseline and after treatment completion about 9 months
  the position of the upper and lower lips, and chin will be measured.
patient acceptance of treatment | After treatment completion about 9 months
  The patient's acceptance to the treatment will be evaluated using a visual analog scale questionnaire after removal of the appliances.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt